CLINICAL TRIAL: NCT06989047
Title: Comparative Study of Preoperative Ultrasound-Guided Pericapsular Nerve Group Block and Femoral Nerve Block for Analgesia Before Spinal Anesthesia in Proximal Femur Fracture Fixation
Brief Title: Ultrasound-Guided PENG Block vs Femoral Nerve Block for Analgesia Before Spinal Anesthesia in Hip Fracture Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Khaled Radwan Ammar, Resident of Anesthesia, Intensive Care and Pain Management, Faculty of Medicine, Ain Shams University, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MS49/2024
Record Dates: First submitted 2025-05-07; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Proximal Femur Fracture; Hip Fracture; Pain Management; Spinal Anesthesia
Keywords: Pericapsular Nerve Group Block (PENG); Femoral Nerve Block (FNB); Ultrasound-Guided Nerve Block; Spinal Anesthesia; Hip Surgery; Regional Anesthesia
MeSH Terms: conditions — Proximal Femoral Fractures; Hip Fractures; Agnosia | interventions — Dental Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG Block Group (Experimental): Assigned Interventions:
  Procedure/Surgery: Pericapsular Nerve Group (PENG) Block An ultrasound-guided nerve block targeting articular branches of the femoral, obturator, and accessory obturator nerves. Performed under aseptic technique using a curved low-frequency ultrasound probe to visualize the iliopsoas plane and pubic ramus.
  Drug: Bupivacaine (0.25%, 30 ml) Local anesthetic used to provide analgesia in nerve block. Drug: Magnesium sulfate (10%, 5 ml = 500 mg) Adjunct used to enhance analgesic efficacy of the block.
  Interventions: Procedure: Pericapsular Nerve Group (PENG) Block
- Femoral Nerve Block Group (Active Comparator): Assigned Interventions:
  Procedure/Surgery: Femoral Nerve Block (FNB) An ultrasound-guided nerve block targeting the femoral nerve, performed with an in-plane ultrasound approach under sterile conditions, identifying the nerve lateral to the femoral artery.
  Drug: Bupivacaine (0.25%, 30 ml) Local anesthetic used for nerve block. Drug: Magnesium sulfate (10%, 5 ml = 500 mg) Adjunct analgesic agent.
  Interventions: Procedure: Femoral Nerve Block (FNB)

INTERVENTIONS:
Procedure: Pericapsular Nerve Group (PENG) Block — Assigned Interventions:
  Procedure/Surgery: Pericapsular Nerve Group (PENG) Block An ultrasound-guided nerve block targeting articular branches of the femoral, obturator, and accessory obturator nerves. Performed under aseptic technique using a curved low-frequency ultrasound probe to visualize the iliopsoas plane and pubic ramus.
  Drug: Bupivacaine (0.25%, 30 ml) Local anesthetic used to provide analgesia in nerve block. Drug: Magnesium sulfate (10%, 5 ml = 500 mg) Adjunct used to enhance analgesic efficacy of the block.
  Arms: PENG Block Group
Procedure: Femoral Nerve Block (FNB) — An ultrasound-guided nerve block targeting the femoral nerve to provide analgesia before spinal anesthesia in proximal femur fracture surgery. Administered using 30 ml of 0.25% bupivacaine and 5 ml of 10% magnesium sulfate (500 mg). The block is performed with an in-plane ultrasound approach, identifying the femoral nerve lateral to the femoral artery under sterile conditions.
  Arms: Femoral Nerve Block Group

SUMMARY:
This study will compare two types of ultrasound-guided nerve blocks-Pericapsular Nerve Group (PENG) block and Femoral Nerve Block (FNB)-to evaluate their effectiveness in reducing pain before spinal anesthesia in patients who will undergo surgery for proximal femur fractures. Proximal femur fractures will continue to be common, especially in older adults, and often will cause severe pain that will make it difficult to position patients for spinal anesthesia. Both nerve blocks will aim to reduce pain, improve comfort during spinal anesthesia, and decrease the need for postoperative pain medication.

A total of 60 adult patients who will undergo proximal femur fracture fixation under spinal anesthesia will be enrolled and randomly assigned to receive either a Pericapsular Nerve Group (PENG) block or a femoral nerve block before the procedure. The study will monitor patients' pain scores using the Visual Analog Scale (VAS) at multiple time points, including during positioning and throughout the first 24 hours after surgery. It also will evaluate how long it will take before the patients require rescue pain medication, and how much total pain medication will be needed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Scheduled for proximal femur fracture fixation under spinal anesthesia
* Classified as American Society of Anesthesiologists (ASA) physical status I, II, or III
* Ability to understand and use the Visual Analog Scale (VAS)
* Provided written informed consent

Exclusion Criteria:

* Coagulopathy
* Local infection at the injection site
* Known allergy to local anesthetics or magnesium sulfate
* Severe cardiopulmonary disease [American Society of Anesthesiologists (ASA) ≥ IV]
* Preexisting diabetic or other neuropathies
* Chronic opioid use
* Contraindication to spinal anesthesia
* Cognitive impairment or inability to comprehend Visual Analog Scale (VAS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-30 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Pain Score During Positioning for Spinal Anesthesia Using Visual Analog Scale (VAS) | Immediately before spinal anesthesia (within 15 minutes post-block)
  The Visual Analog Scale (VAS) will be used to assess pain intensity during positioning for spinal anesthesia. The VAS is a 10 cm line where 0 indicates no pain and 10 indicates the worst imaginable pain. The score will be recorded immediately before spinal anesthesia after performing either the PENG block or femoral nerve block.
Time to First Rescue Analgesia | Within 24 hours postoperatively
  The time (in hours) from the end of the nerve block to the first request for additional analgesia (nalbuphine 0.2 mg/kg IV) will be recorded for each patient.

SECONDARY OUTCOMES:
Total Nalbuphine Consumption | 24 hours postoperatively
  The cumulative dose (in mg) of intravenous nalbuphine administered for pain control will be calculated for each participant over the first 24 hours following surgery.
Mean Arterial Pressure (MAP) Changes | From baseline up to 24 hours postoperatively
  Mean arterial pressure will be recorded at baseline (pre-block), then at 2, 5, 10, 15 minutes post-block, and subsequently at 2, 6, 12, 18, and 24 hours after surgery to evaluate hemodynamic stability following either pericapsular nerve block (PENG) block or femoral nerve block.
Patient Satisfaction Score | At 24 hours postoperatively
  Patient satisfaction with pain control will be evaluated using a 5-point Likert scale (1 = very dissatisfied, 5 = very satisfied) at the end of the 24-hour postoperative period.

IPD SHARING:
Plan to Share IPD: No